CLINICAL TRIAL: NCT03298984
Title: A Phase 1, Open-label, Dose-escalation, Safety and Biomarker Prediction of Alvocidib and Cytarabine/Daunorubicin (7+3) in Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Brief Title: Ph I Study of Alvocidib and Cytarabine/Daunorubicin (7+3) in Patients With Newly Diagnosed Acute Myeloid Leukemia (AML).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPI-ALV-101
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Results first posted 2021-05-24 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — alvocidib; Cytarabine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alvocidib and Cytarabine/Daunorubicin (Experimental): The starting dose of alvocidib will be 20 mg/m2 as a 30-minute intravenous (IV) bolus followed by 30 mg/m2 over 4 hours as an IV infusion administered daily on Days 1-3 of Induction. Patients will have a one day drug holiday (Day 4) before initiation of the 7+3 regimen. Beginning on Day 5, cytarabine will be administered as a 100 mg/m2/day continuous IV infusion for seven consecutive days (Days 5-11) plus daunorubicin administered at a dosage of 60 mg/m2 IV on Days 5-7.
  Interventions: Drug: Alvocidib; Drug: Cytarabine; Drug: Daunorubicin

INTERVENTIONS:
Drug: Alvocidib — IV bolus followed by IV infusion
Drug: Cytarabine — continuous infusion
Drug: Daunorubicin — IV bolus

SUMMARY:
The purpose of this Phase I study is to determine the safety and tolerability including the maximum dose (MTD) and dose-limiting toxicities (DLTs) of alvocidib when administered over a range of doses on Days 1-3 followed by cytarabine/daunorubicin (7+3) on Days 5-11 in adults with newly diagnosed and previously untreated AML

DETAILED DESCRIPTION:
Primary Objective:

• To determine the safety and tolerability including the maximum tolerated dose (MTD) and dose-limiting toxicities (DLTs) of alvocidib when administered over a range of doses on Days 1-3 followed by cytarabine/daunorubicin (7+3) on Days 5-11 in adults with newly diagnosed and previously untreated AML

Secondary Objectives:

* To observe patients for any evidence of antileukemic activity of alvocidib plus 7+3 using the 2017 ELN response criteria
* To establish the Recommended Phase 2 Dose (RP2D) for future studies with alvocidib in combination with 7+3

Exploratory Objective:

• To assess levels of minimal residual disease (MRD) using standardized techniques (ie, multiparametric flow cytometry [MPFC] and next generation sequencing [NGS] and evaluate other potential biomarkers including, but not limited to, MCL-1 dependency.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for participation in the study, patients must meet all of the following inclusion criteria:

  1. Be between the ages of ≥18 and ≤65 years
  2. Have an established, pathologically confirmed diagnoses of AML by World Health Organization (WHO) criteria with ≥20% bone marrow blasts based on histology or flow cytometry
  3. Be newly diagnosed and previously untreated
  4. Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤2
  5. Have a serum creatinine level ≤1.8 mg/dL
  6. Have an alanine aminotransferase (ALT) and aspartate aminotransferase (AST) level ≤5 times upper limit of normal (ULN)
  7. Have a total bilirubin level ≤2.0 mg/dL (unless secondary to Gilbert syndrome, hemolysis, or leukemia)
  8. Have a left ventricular ejection fraction (LVEF) >45% by echocardiogram (ECHO) or multigated acquisition (MUGA) scan
  9. Be nonfertile or agree to use an adequate method of contraception. Sexually active patients and their partners must use an effective method of contraception associated with a low failure rate prior to study entry, for the duration of study participation, and for at least 6 months after the last dose of study drug.
  10. Be able to comply with the requirements of the entire study.
  11. Provide written informed consent prior to any study related procedure. (In the event that the patient is re-screened for study participation or a protocol amendment alters the care of an ongoing patient, a new informed consent form must be signed.)

Exclusion Criteria:

* Patients meeting any one of these exclusion criteria will be prohibited from participating in this study.

  1. Received any previous treatment for AML
  2. Diagnosed with APL-M3 or CBF-AML
  3. Require concomitant chemotherapy, radiation therapy, or immunotherapy. Hydroxyurea is allowed up to the evening before starting (but not within 12 hours) of starting Induction therapy.
  4. Received >200 mg/m2 equivalents of daunorubicin
  5. Have a peripheral blast count of >30,000/mm3 (may use hydroxyurea as in #3 above)
  6. Have active central nervous system (CNS) leukemia
  7. Have evidence of uncontrolled disseminated intravascular coagulation
  8. Have an active, uncontrolled infection
  9. Have other life-threatening illness
  10. Have other active malignancies or diagnosed with other malignancies within the last 6 months, except nonmelanoma skin cancer or cervical intraepithelial neoplasia
  11. Have mental deficits and/or psychiatric history that may compromise the ability to give written informed consent or to comply with the study protocol.
  12. Are pregnant and/or nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Anthony, DO, Study Director — Sumitomo Pharma America, Inc.
Locations (3):
- United States (3):
  - Sidney Kimmel Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Columbia University, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zeidner JF, Lee DJ, Frattini M, Fine GD, Costas J, Kolibaba K, Anthony SP, Bearss D, Smith BD. Phase I Study of Alvocidib Followed by 7+3 (Cytarabine + Daunorubicin) in Newly Diagnosed Acute Myeloid Leukemia. Clin Cancer Res. 2021 Jan 1;27(1):60-69. doi: 10.1158/1078-0432.CCR-20-2649. Epub 2020 Sep 30. PMID 32998965

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 32 patients at 3 sites; Recruitment started 25Sep2017 Recruitment ended 20Mar2020
Pre-assignment Details: 4 dose escalation cohorts. If 1 of 3 subjects in a cohort experienced a DLT, up to 3 additional subjects were treated at that dose level. If no DLTs observed, the alvocidib dose was escalated in a new cohort of 3 subjects. At MTD level 20 additional subjects enrolled for confirmation of safety as well as additional safety analysis.
Groups:
- Alvocidib 20/30 mg/m2: Alvocidib 20 mg/m2 bolus followed by 30 mg/m2 IV infusion over 4 hours
- Alvocidib 30/40 mg/m2: Alvocidib 30 mg/m2 bolus followed by 40 mg/m2 IV infusion over 4 hours
- Alvocidib 30/50 mg/m2: Alvocidib 30 mg/m2 bolus followed by 50 mg/m2 IV infusion over 4 hours
- Alvocidib 30/60 mg/m2: Alvocidib 30 mg/m2 bolus followed by 60 mg/m2 IV infusion over 4 hours
Period: Overall Study
Arm/Group | Alvocidib 20/30 mg/m2 | Alvocidib 30/40 mg/m2 | Alvocidib 30/50 mg/m2 | Alvocidib 30/60 mg/m2
Started | 3 | 3 | 3 | 23
Completed | 2 | 2 | 1 | 8
Not Completed | 1 | 1 | 2 | 15
Not completed — Physician Decision | 1 | 0 | 0 | 6
Not completed — Lack of Efficacy | 0 | 1 | 1 | 4
Not completed — Relapsed disease (following remission) | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 2
Not completed — Insurance Company Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alvocidib 20/30 mg/m2 | Alvocidib 30/40 mg/m2 | Alvocidib 30/50 mg/m2 | Alvocidib 30/60 mg/m2 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 23 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 23 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 9 | 14
  Male | 1 | 1 | 2 | 14 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 2 | 5
  White | 1 | 1 | 2 | 20 | 24
  More than one race | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Alvocidib
Description: Determine the safety and tolerability including the maximum tolerated dose (MTD) of alvocidib when administered over a range of doses on Days 1-3 followed by Ara-c/daunorubicin (7+3) on Days 5-11 in adults with newly diagnosed and previously untreated AML
Time Frame: During the first cycle
Measure: Number; unit: mg/m2
Groups:
- All Participants: All participants who received at least 1 dose of Alvocidib, either at 20 mg/m2 bolus followed by 30 mg/m2 IV infusion over 4 hours, 30 mg/m2 bolus followed by 40 mg/m2 IV infusion over 4 hours, 30 mg/m2 bolus followed by 50 mg/m2 IV infusion over 4 hours, or 30 mg/m2 bolus followed by 60 mg/m2 IV infusion over 4 hours
Arm/Group | All Participants
Number analyzed (Participants) | 32
mg/m2
  Bolus | 30
  IV infusion | 60

2. Primary Outcome: Number of Participants Who Experienced Dose Limiting Toxicities (DLTs) of Alvocidib
Description: Determine the safety and tolerability including dose-limiting toxicities (DLTs) of alvocidib when administered over a range of doses on Days 1-3 followed by Ara-c/daunorubicin (7+3) on Days 5-11 in adults with newly diagnosed and previously untreated AML
Time Frame: During the first cycle
Measure: Count of Participants; unit: Participants
Arm/Group | Alvocidib 20/30 mg/m2 | Alvocidib 30/40 mg/m2 | Alvocidib 30/50 mg/m2 | Alvocidib 30/60 mg/m2
Number analyzed (Participants) | 3 | 3 | 3 | 23
Participants | 0 | 0 | 0 | 1

3. Secondary Outcome: Antileukemic Activity of Alvocidib Plus 7+3 - Response to Treatment Based on 2017 ELN Response Criteria
Description: CR: Measurable residual disease is positive or unknown; BM blasts (bls) <5%; no circulating bls and bls w/ Auer rods; no extramedullary disease; ANC >1.0 x 109/L; platelets >100 x 109/L. CRMRD-: CR w/ negativity genetic marker. CRi: CR except residual neutropenia or thrombocytopenia. MLFS: BM bls <5%; no bls with Auer rods; no extramedullary disease; no hematologic recovery required. PR: all hematologic CR criteria; decrease (dec) BM bls % to 5-25%; dec pretreatment BM bls % by >50%. SD: no CRMRD-/CR/CRi/PR/MLFS; PD criteria not met. PD: increase (inc) BM bls % and/or inc absolute bls in blood: 50% inc BM bls over baseline (>15% point inc required in cases w/ <30% bls at baseline or persistent BM bls % of >70% over at least 3 months; without at least 100% improvement in ANC to absolute level [>0.5 x 109/L and/or platelet count to >50 x 109/L non-transfused); or >50% inc in peripheral bls to >25 x 109/L (in the absence of differentiation syndrome); or new extramedullary disease.
Time Frame: Best response during duration of study
Measure: Number; unit: participants
Arm/Group | Alvocidib 20/30 mg/m2 | Alvocidib 30/40 mg/m2 | Alvocidib 30/50 mg/m2 | Alvocidib 30/60 mg/m2
Number analyzed (Participants) | 3 | 3 | 3 | 23
participants
  Complete Remission MRD Negative (CRMRD-) | 2 | 0 | 2 | 8
  Complete Remission MRD Positive or Unknown (CR) | 1 | 2 | 0 | 7
  Partial Remission (PR) | 0 | 1 | 0 | 1
  Stable Disease | 0 | 0 | 0 | 2
  Progressive Disease (PD) | 0 | 0 | 1 | 4
  Not Evaluated | 0 | 0 | 0 | 1

4. Secondary Outcome: Recommended Phase 2 Dose (RP2D) of Alvocidib in Combination With 7+3
Description: The dose at which < 1 of 6 patients experience a DLT during Cycle 1 with the next higher dose having at least 2 of 3 to 6 patients experiencing a DLT during Cycle 1
Time Frame: During Cycle 1 beginning at 1st dose of study drug through Day 50 + or - 3 days
Measure: Number; unit: mg/m2
Arm/Group | All Participants
Number analyzed (Participants) | 32
mg/m2
  Bolus | 30
  IV infusion | 60

5. Other Pre Specified Outcome: Minimal Residual Disease (MRD) Using Standardized Techniques
Description: Percentage of participants with a CRMRD- response at the end of Cycle 1
Time Frame: During duration of study
Measure: Number; unit: percentage of participants
Arm/Group | Alvocidib 20/30 mg/m2 | Alvocidib 30/40 mg/m2 | Alvocidib 30/50 mg/m2 | Alvocidib 30/60 mg/m2
Number analyzed (Participants) | 3 | 3 | 3 | 23
percentage of participants | 66.7 | 0 | 66.7 | 34.8

ADVERSE EVENTS:
Time Frame: Beginning at 1st dose of study drug through 30 days of the last administration of study drug
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Groups:
- Alvocidib 20/30 mg/m2 (N=3): Alvocidib 20mg/m2 bolus followed by 30 mg/m2 IV infusion over 4 hours
- Alvocidib 30/40 mg/m2 (N=3): Alvocidib 30 mg/m2 bolus followed by 40 mg/m2 IV infusion over 4 hours
- Alvocidib 30/50 mg/m2 (N=3): Alvocidib 30 mg/m2 bolus followed by 50 mg/m2 IV infusion over 4 hours
- Alvocidib 30/60 mg/m2 (N=23): Alvocidib 30 mg/m2 bolus followed by 60 mg/m2 IV infusion over 4 hours
Arm/Group | Alvocidib 20/30 mg/m2 (N=3) | Alvocidib 30/40 mg/m2 (N=3) | Alvocidib 30/50 mg/m2 (N=3) | Alvocidib 30/60 mg/m2 (N=23)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 2/23
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/3 | 5/23
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alvocidib 20/30 mg/m2 (N=3) (N=3) | Alvocidib 30/40 mg/m2 (N=3) (N=3) | Alvocidib 30/50 mg/m2 (N=3) (N=3) | Alvocidib 30/60 mg/m2 (N=23) (N=23)
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1
Fungaemia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alvocidib 20/30 mg/m2 (N=3) (N=3) | Alvocidib 30/40 mg/m2 (N=3) (N=3) | Alvocidib 30/50 mg/m2 (N=3) (N=3) | Alvocidib 30/60 mg/m2 (N=23) (N=23)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 3 | 19
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 4
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 7
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 2
Keratitis (Eye disorders) | 1 | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 1 | 0 | 1
Eye inflammation (Eye disorders) | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 3 | 23
Nausea (Gastrointestinal disorders) | 1 | 2 | 2 | 17
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 14
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 10
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 6
Constipation (Gastrointestinal disorders) | 0 | 2 | 3 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 5
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1 | 5
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 4
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 2 | 12
Fatigue (General disorders) | 2 | 2 | 1 | 8
Chills (General disorders) | 1 | 0 | 1 | 4
Pyrexia (General disorders) | 1 | 1 | 0 | 4
Catheter site pain (General disorders) | 0 | 0 | 1 | 3
Chest pain (General disorders) | 0 | 1 | 0 | 3
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 3
Oedema (General disorders) | 0 | 0 | 0 | 2
Pain (General disorders) | 0 | 0 | 0 | 2
Localised oedema (General disorders) | 0 | 0 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 2 | 7
Lung infection (Infections and infestations) | 0 | 2 | 0 | 4
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 2
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2
Bacteraemia (Infections and infestations) | 2 | 0 | 1 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 1
Enterococcal infection (Infections and infestations) | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Abdominal infection (Infections and infestations) | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis orbital (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 1 | 0 | 0 | 0
Fungaemia (Infections and infestations) | 1 | 0 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 1 | 0 | 0 | 0
Oral infection (Infections and infestations) | 0 | 1 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 4
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lip injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 2 | 2 | 9
Platelet count decreased (Investigations) | 0 | 1 | 2 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 3 | 3
Blood bilirubin increased (Investigations) | 0 | 1 | 2 | 3
Blood creatinine increased (Investigations) | 1 | 2 | 1 | 3
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 3
Lymphocyte count decreased (Investigations) | 0 | 1 | 2 | 3
Weight decreased (Investigations) | 1 | 1 | 0 | 3
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 1
Neutrophil count decreased (Investigations) | 2 | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0
Sputum culture positive (Investigations) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2 | 3 | 16
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 10
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0 | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 5
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 3
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Cytarabine syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 1 | 10
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 8
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 2
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 6
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 3
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 1 | 4
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 4
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 7
Hypertension (Vascular disorders) | 0 | 0 | 1 | 3
Embolism (Vascular disorders) | 0 | 0 | 0 | 2
Flushing (Vascular disorders) | 0 | 0 | 1 | 1
Jugular vein distension (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT03298984/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT03298984/SAP_001.pdf